CLINICAL TRIAL: NCT05284045
Title: Study of the Nocebo Effect in Patients With Obstructive Sleep Apnea Syndrome and Treatment With Continuous Positive Airway Pressure
Brief Title: Nocebo Effect in OSA Patients With CPAP Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Mireia Dalmases, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HCB/2021/1330
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual information (No Intervention): Subjects allocated to this arm will receive the usual information about OSA and CPAP treatment given in clinical practise
- Detailed information (Active Comparator): Subjects allocated to this arm will also receive the usual information about OSA and CPAP treatment and they will also receive information related to the possible adverse side effects of CPAP treatment. The healthcare professional will enumerate the possible side effects and indicate which are more and less common.
  Interventions: Other: Detailed information

INTERVENTIONS:
Other: Detailed information — Subjects in this arm will receive usual information + detailed information on side effects
  Arms: Detailed information

SUMMARY:
This study is aimed to evaluate whether the information provided by health care professionals in the visits previous to start with CPAP treatment may influence the number of reported adverse effects and compliance in patients with obstructive sleep apnea (OSA) in treatment with CPAP.

DETAILED DESCRIPTION:
Background: The presence of side effects in the first few weeks of treatment with CPAP is common. However, it has never been evaluated whether side effects could be related to the presence of the nocebo effect in this population.

Main objective: To assess whether the information provided by health care professionals may influence the number of reported adverse events and compliance in patients with obstructive sleep apnea (OSA) in treatment with CPAP.

Methodology: Unicentric randomized clinical trial that will include 80 patients over 18 years of age with a recent diagnosis of OSA and indication for treatment with CPAP. Participants will be recruited consecutively and will be randomly assigned in a 1: 1 ratio to receive usual information or more detailed information in possible adverse effects of treatment during the CPAP adaptation visit. Follow-up will be performed at 1 month and 3 months after starting CPAP treatment. Side effects and treatment compliance in each of the groups will be blindly assessed. Descriptive statistics and differences in the number of side effects and hours of compliance between the two groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with OSA with indication for CPAP treatment
2. To be over 18 years old
3. Sign informed consent for study participation.

Exclusion Criteria:

1. Patients previously treated with CPAP.
2. Patients with other previous treatments for OSA (surgery, mandibular advancement device, etc.)
3. Presence of any other previously diagnosed sleep disorder
4. Patients with> 50% central sleep apnea or Cheyne-Stokes respiration
5. Diagnosis of a mental or physical condition that makes difficult to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Number of side effects | at 1 month
  Evaluate the number of side effects reported in both arms

SECONDARY OUTCOMES:
Hours of CPAP use | at 3 month
  Number of hours will be collected from the internal clock of the CPAP device

CONTACTS AND LOCATIONS:
Overall Officials: Mireia DALMASES CLERIES, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain